CLINICAL TRIAL: NCT05424718
Title: MyPEEPS (Male Youth Pursuing Empowerment, Education, and Prevention Around Sexuality) Mobile for Young Transgender Men
Brief Title: MyPEEPS Mobile for Young Transgender Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Callen-Lorde Community Health Center (Other)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT8624; R34MH128163 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: HIV
Keywords: MyPEEPS; Mobile Intervention; Human Immunodeficiency Virus (HIV); Transgender Youth
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The intervention arm receives the intervention from baseline to 3 months and at the 3 month visit, access to the intervention is removed and the control/ delayed intervention arm then receives the intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Study participants randomized to the intervention arm will have access to the MyPEEPS Mobile application for the first three months of the trial and then the intervention is removed at the 3 month follow-up visit.
  Interventions: Behavioral: MyPEEPS Mobile
- Delayed Intervention (Experimental): Participants randomized to the delayed intervention arm will not have access to MyPEEPS Mobile for the first 3 months of the study and will receive access to the MyPEEPS Mobile App at the 3 month follow-up visit.
  Interventions: Behavioral: MyPEEPS Mobile

INTERVENTIONS:
Behavioral: MyPEEPS Mobile — Mobile technology to deliver HIV prevention information specifically developed for at-risk young men that have sex with men (YMSM).

SUMMARY:
The proposed MyPEEPS intervention for young transgender men is a novel and evidence-driven intervention using mobile technology to deliver HIV prevention information to high risk youth. The final product will be the basis for conducting a large-scale efficacy study in this population.

DETAILED DESCRIPTION:
Transgender youth in the United States have unique health needs but often face barriers to accessing and receiving health care services which contribute to disparate health outcomes including high vulnerability to HIV and other sexually transmitted infections. Emerging evidence has begun to document HIV-related sexual risk among young transgender men (YTM), as well as low uptake of pre-exposure prophylaxis among those with indications, suggesting high vulnerability to HIV infection. Despite the high prevalence and increased risk of HIV in YTM who have sex with cisgender men, only one prior HIV prevention intervention has been developed to address the specific sexual health needs of YTM, which indicates a critical gap in HIV prevention science. In response to this need, and building off preliminary work, the investigators propose to develop a mobile intervention for YTM building on MyPEEPS Mobile, which was originally developed for very young sexual minority men. Central to this intervention is the premise that it will be delivered to youth during a developmental period that precedes or coincides with sexual debut, an important time for intervention, prior to or concurrent with initiation of high-risk behaviors.

Given both the gap in HIV prevention science and the lack of current targeted interventions, and building upon our multidisciplinary team's extensive experience in HIV prevention, mobile health (mHealth), behavioral interventions, randomized controlled trials, and transgender health, the investigators propose the following specific aims: 1) Using qualitative methodology, expert feedback, and usability assessments, develop MyPEEPS Mobile for YTM, 2) Conduct a pilot randomized controlled trial to examine the feasibility, acceptability, and preliminary efficacy of the revised MyPEEPS Mobile App in a sample of 80 YTM (15-25 years) and refine the study methods for a future efficacy trial, and 3) Assess predisposing, enabling, and reinforcing factors for MyPEEPS Mobile among YTM through theoretically-guided in depth interviews. The proposed MyPEEPS intervention for YTM will be the first study to develop and pilot a scaled-up, mobile HIV prevention intervention designed by, and piloted for, a diverse group of YTM. The final product of this study will be the basis for an R01 application to conduct a large-scale efficacy study for this population.

ELIGIBILITY:
Inclusion Criteria:

To participate in any aspect of the study, participants must be:

* Between 15 and 25 years of age;
* Female sex assigned at birth;
* Identify as a transgender man or along the transmasculine spectrum (including a transmasculine non-binary gender; e.g., male, trans male, transmasculine gender non-binary);
* Understand and read English;
* Live within the US;
* Own a smartphone;
* Self-report condomless receptive anal or vaginal penile sex with either a cisgender male or transgender woman (e.g., individual designated or assigned male at birth) in the past year; and
* Self-report HIV-negative or unknown status.

Exclusion Criteria:

Youth are ineligible to participate in the trial if:

* HIV positive;
* Unable to provide informed consent due to severe mental or physical illness or substance intoxication at the time of enrollment;
* Concurrently enrolled in another HIV prevention study.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Identify as a transgender man or along the transmasculine spectrum (including a transmasculine non-binary gender; e.g., male, trans male, transmasculine gender non-binary);
Enrollment: 80 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Ann & Robert H. Lurie Children's Hospital Chicago, Chicago, Illinois
  - Callen-Lorde Community Health Center, New York, New York
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No
While individual participant data (IPD) will not be shared, the results of the study will be shared at conferences such as the American Public Health Association annual meeting and Infectious Disease week; provide organizations that are influential in HIV public health practice (e.g., International AIDS Society) with an executive summary, press releases, and/or published papers; publish results in peer-reviewed academic journals; provide a lay summary for participants and community partners.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Intervention | Delayed Intervention
Started | 40 | 40
Completed | 35 | 36
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Delayed Intervention | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (2.4) | 22.2 (2.4) | 22 (2.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transgender Man | 14 | 14 | 28
  Non-binary | 9 | 3 | 12
  Other | 17 | 23 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 11 | 13 | 24
  White | 17 | 12 | 29
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Self-Reported Nonoccupational Human Immunodeficiency Virus (HIV) Postexposure Prophylaxis (nPEP) Use [Number; unit: participants] — The number of participants that self-reported Nonoccupational HIV Postexposure Prophylaxis (nPEP) use.
  participants | 0 | 3 | 3
Self-reported Pre-exposure Prophylaxis (PrEP) Use [Count of Participants; unit: Participants] — Number of participants that self-reported Pre-exposure Prophylaxis (PrEP) Use
  Participants | 6 | 7 | 13
Self-reported HIV Testing [Count of Participants; unit: Participants] — Number of participants that self-reported HIV testing
  Participants | 18 | 16 | 34
Self-reported Sexually Transmitted Infection (STI) Testing [Number; unit: participants] — Number of participants that self-reported STI testing
  participants | 25 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Condomless Receptive Sex Acts
Description: Change in self-reported number of condomless receptive anal or vaginal sex acts with sex partners assigned male at birth
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: Condomless Receptive Sex Acts
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 35 | 36
Condomless Receptive Sex Acts
  Baseline and 3 Months | 1.57 (5.55) | 3.19 (9.75)
  3 Months and 6 Months | 1.43 (6.4) | 1.44 (17.7)

2. Secondary Outcome: Self-reported Nonoccupational HIV Postexposure Prophylaxis (nPEP) Use
Description: Number of participants that self-reported nPEP use
Time Frame: 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 35 | 36
Participants
  3 months | 1 | 2
  6 months | 1 | 4

3. Secondary Outcome: Self-reported Pre-exposure Prophylaxis (PrEP) Use
Description: Number of participants that self-reported Pre-exposure Prophylaxis (PrEP) Use
Time Frame: 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 35 | 36
Participants
  3 Months | 6 | 7
  6 Months | 6 | 7

4. Secondary Outcome: Self-reported HIV Testing
Description: Number of participants that self-reported HIV testing
Time Frame: 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 35 | 36
Participants
  3 Months | 12 | 21
  6 Months | 15 | 17

5. Secondary Outcome: Self-reported Sexually Transmitted Infections (STI) Testing
Description: Number of participants that self-reported STI Testing
Time Frame: 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 35 | 36
Participants
  3 Months | 19 | 23
  6 Months | 19 | 20

6. Secondary Outcome: Change in Partner PrEP Use and Adherence or Viral Suppression
Description: Change in participant's self-report of their partner(s) PrEP use and adherence or viral suppression (if partner(s) is HIV+)
Time Frame: Baseline, 3 and 6 months
Population: Data was not analyzed as participant's self-report of partner(s) PrEP use and adherence/viral supression data were not collected (due to unintentional omision of partner related questions in the participant questionnaire).
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Immediate Intervention | Delayed Intervention
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any presentation, abstract, or manuscript will be made available for review by the study sponsor(s) prior to submission

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT05424718/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT05424718/ICF_001.pdf